CLINICAL TRIAL: NCT07116187
Title: A Pilot Return-to-Work Cognitive Intervention After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Catherine Yanhong Dong, PhD, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: NUS-IRB-2025-223
Record Dates: First submitted 2025-07-22; First posted 2025-08-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Cognition; Return-to-work; Rehabilitation; Intervention; Community; Stroke survivors; Caregivers
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants will undergo the group-based Train-Your-Brain Stroke Recovery Programme.
  Interventions: Other: Train-Your-Brain (TYB) Stroke Recovery Programme
- Control Arm (No Intervention): Participants will undergo treatment-as-usual from their respective treatment providers.

INTERVENTIONS:
Other: Train-Your-Brain (TYB) Stroke Recovery Programme — The intervention involves a structured brain health programme delivered by clinical neuropsychologists in three phases: an initial needs assessment, a multi-session intervention, and follow-up support. Participants will receive assessments, attend group sessions covering topics such as lifestyle, mood, cognition, and return-to-work strategies, and be supported with workbooks and referrals to community services. The programme combines in-person and online formats.
  Arms: Intervention Arm

SUMMARY:
This study addresses the growing burden of stroke in Singapore and highlights the lack of rehabilitation services for return to work after stroke. Despite functional physical recovery, many stroke survivors experience persistent impairments that hinder return-to-work. To bridge this gap, the study will implement a community-based brain health programme targeting cognitive and vocational outcomes in stroke survivors. Caregivers will also be included due to their critical support role. The study will assess the intervention's feasibility, acceptability, and its impact on cognitive function, return-to-work, neuroplasticity, psychosocial health, fatigue, and self-care.

DETAILED DESCRIPTION:
Stroke is the fourth leading cause of death and the leading cause of adult disability in Singapore. Statistics indicate a concerning rise in young stroke cases. The burden of stroke care is expected to increase exponentially, posing significant challenges to the healthcare system and society. Cognitive impairment after stroke has been documented in up to one-third of stroke survivors. These impairments may be subtle but persistent and progressive even after the stroke survivor appears to have made functional recovery in other areas. Existing services in Singapore for stroke survivors typically target physical and daily functioning outcomes with little focus on cognitive functioning. Moreover, there is a lack of services for stroke survivors who face difficulties in returning to work due to cognitive impairment even when they have achieved optimal physical recovery. An important assessment of a rehabilitation intervention programme is in examining whether it drives positive neuroplasticity, which leads to improved cognitive and functional outcomes. There is presently a dearth of literature in brain mechanisms underlying the impact of cognitive rehabilitation.

A community-based brain health intervention, the Train-Your-Brain Stroke Recovery Programme, will be delivered by registered clinical neuropsychologists. Designed to enhance cognitive function and return-to-work outcomes in stroke survivors with mild cognitive impairment, the intervention will be evaluated using a mixed-methods randomized controlled trial. Stroke survivors will be randomized 1:1 into either the intervention or control arm. Caregivers, given their critical support role, will also be recruited to participate in the study. Outcome measures include feasibility of intervention, acceptability of intervention, cognitive function, return-to-work outcomes, changes in biomarkers, neuroimaging findings, psychosocial health, fatigue, and self-care. Outcome measures will be conducted pre-intervention, post-intervention, and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria (for stroke survivors):

* Between 21 to 65 years old
* Ability to provide informed consent
* Consent to recording / photo-taking
* Living in the community with at least three months after stroke
* Looking to return to work or switch jobs after stroke
* No significant aphasia or physical disability issues which will impede them from performing cognitive tasks in the interventions and assessments
* No major psychiatric illnesses
* Able to understand and converse in English
* Score on MoCA ≤22 and/or SDMT ≤13 (for those educated ≤6 years) or SDMT ≤32 (for those educated >6 years)
* Meet criteria for Mild Cognitive Impairment based on the Vascular Dementia Battery

Inclusion Criteria (for caregivers):

* At least 21 years old
* Ability to provide informed consent
* Consent to recording / photo-taking
* Staying with or having knowledge of the stroke survivor's functioning
* No major psychiatric illnesses
* Able to understand and converse in English

Exclusion Criteria (for stroke survivors):

* Less than 21 years old
* More than 65 years old
* Unable to provide informed consent
* Refuse recording
* Not living in the community and having less than three months after stroke
* Significant aphasia or physical disability issues which will impede them from performing cognitive tasks in the interventions and assessments
* Major psychiatric illnesses
* Not able to understand and converse in English

Exclusion Criteria (for caregivers):

* Less than 21 years old
* Unable to provide informed consent
* Refuse recording
* Not staying with or not having knowledge of the stroke survivor's functioning
* Major psychiatric illnesses
* Not able to understand and converse in English

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of eligible/ineligible participants | Through study completion, an average of 6 months
  Percentage of eligible/ineligible participants and reasons for ineligibility
Recruitment and attrition rates | Through study completion, an average of 6 months
  Percentage of recruited participants and drop-outs
VasCog Screen Test | Baseline (pre-intervention), immediately after the intervention, 6-months follow-up
  Test is comprised of a short-Montreal Cognitive Assessment (total score out of 12) and modified Symbol Digit Modalities Test (score calculated based on correct responses)
Vascular Dementia Battery | Baseline (pre-intervention)
  Participants will meet criteria for Mild Cognitive Impairment if there is 1 or more domain(s) with failure in at least 50% of tasks in domain
National Institute of Neurological Disorders and Stroke - Canadian Stroke Network (NINDS-CSN) Stroke Protocol | Baseline (pre-intervention), immediately after the intervention, 6-months follow-up
  A test battery comprised of cognitive tests that are measured against their respective normative scores
Return-to-work Questionnaire (National Institute of Neurological Disorders and Stroke - Common Data Elements) | Baseline (pre-intervention), immediately after the intervention, 6-months follow-up
  Survey questions of participants' work status before and after stroke with check-box responses
Intervention fidelity | During the intervention and immediately after the intervention
  Intervention Fidelity Checklist (eNACT Group Facilitation Competency Checklist)
  * "Observed - Done well" and "Observed - Done adequately" is equivalent to a score of 2; "Observed - Not done well" is equivalent to a score of 1; "Not observed - despite opportunity" is equivalent to a score of 0
  * An overall score of 2 reflects adequate competence in group facilitation
Qualitative interviews | Immediately after the intervention
  Semi-structured interviews will be conducted with stroke survivors and family members to obtain feedback about their experiences of the intervention
Participants' acceptability of the intervention | During the intervention
  Feedback forms provided after each intervention session rated on a 5-point response scale from Strongly Disagree to Strongly Agree
Patient-Reported Outcomes Measurement Information System (PROMIS) - 10 | Baseline (pre-intervention), immediately after the intervention, 6-months follow-up
  5-point response scale from Excellent (5) to Poor (1)
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | Baseline (pre-intervention), immediately after the intervention, 6-months follow-up
  Survey questions of participants' Mobility, Self-care, Usual activities, Pain/discomfort, and Anxiety/depression with check-box responses across five levels of severity, ranging from no problems to extreme problems.
Fatigue Assessment Scale | Baseline (pre-intervention), immediately after the intervention, 6-months follow-up
  5-point response scale from Always (5) to Never (1)
Depression, Anxiety, Stress Scale | Baseline (pre-intervention), immediately after the intervention, 6-months follow-up
  3-point response scale from Did not apply to me at all (0) to Applied to me very much, or most of the time (3)
Zarit Burden Interview | Baseline (pre-intervention), immediately after the intervention, 6-months follow-up
  4-point response scale from Nearly Always (4) to Never (0)
Voils Domains Of Subjective Extent of Nonadherence | Baseline (pre-intervention), immediately after the intervention, 6-months follow-up
  Survey questions on participants' extent and reasons for nonadherence with check-box responses (None of the time, A little of the time, Some of the time, Most of the time, Every time)
Blood Pressure Measurement | Baseline (pre-intervention), immediately after the intervention, 6-months follow-up
  Measurement of participants' blood pressure reading
Blood-Derived Neurotrophic Factor | Immediately after the intervention, 6-months follow-up
  Blood biomarker derived from participants' blood samples
Functional near-infrared spectroscopy measurement | Immediately after the intervention, 6-months follow-up
  Measurement of oxyhaemoglobin (HbO2), deoxyheemoglobin (HbR), and regional oxygen saturation (rSO2) while participants undergo various cognitive tests (e.g. N-back Task, verbal fluency test, Stroop Task)

SECONDARY OUTCOMES:
Cost Effectiveness Analysis Questionnaire | Immediately after the intervention, 6-months follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
All collected and deidentified IPD